CLINICAL TRIAL: NCT00402350
Title: Safety, Tolerability, and Pharmacokinetics of Staccato® Fentanyl for Inhalation in Normal, Healthy Volunteers
Brief Title: Staccato Fentanyl Single and Multidose PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-003-101; 8 May 2006
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2008-02

CONDITIONS: Breakthrough Pain
Keywords: Staccato Fentanyl, Pharmacokinetics, Pharmacodynamics, inhaled fentanyl
MeSH Terms: conditions — Breakthrough Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator): Subjects (2) from each of the 4 dose escalation arms
  Interventions: Drug: Inhaled Placebo
- 25 mcg IV and Inhaled Crossover (Experimental): Single dose crossover (IV vs Inhaled)
  Interventions: Drug: Inhaled Fentanyl 25 mcg; Drug: Intravenous Fentanyl 25 mcg
- Inhaled fentanyl 25 mcg x 2 (Experimental): Inhaled Staccato fentanyl, 25 mcg x 2
  Interventions: Drug: Inhaled Fentanyl 25 mcg x 2
- Inhaled fentanyl 25 mcg x 4 (Experimental): Inhaled Staccato fentanyl, 25 mcg x 4
  Interventions: Drug: Inhaled Fentanyl 25 mcg x 4
- Inhaled fentanyl 25 mcg x 6 (Experimental): Inhaled Staccato fentanyl, 25 mcg x 6
  Interventions: Drug: Inhaled Fentanyl 25 mcg x 6
- Inhaled fentanyl 25 mcg x 12 (Experimental): Inhaled Staccato fentanyl, 25 mcg x 12
  Interventions: Drug: Inhaled Fentanyl 25 mcg x 12

INTERVENTIONS:
Drug: Inhaled Placebo — Inhaled Staccato Placebo, same number of doses as active comparator in that arm
  Arms: Placebo
Drug: Inhaled Fentanyl 25 mcg — Inhaled Staccato Fentanyl, 25 mcg x 1 dose
  Arms: 25 mcg IV and Inhaled Crossover
Drug: Intravenous Fentanyl 25 mcg — Intravenous Fentanyl 25 mcg, single dose
  Arms: 25 mcg IV and Inhaled Crossover
Drug: Inhaled Fentanyl 25 mcg x 2 — Inhaled Staccato Fentanyl, 25 mcg x 2 doses
  Arms: Inhaled fentanyl 25 mcg x 2
Drug: Inhaled Fentanyl 25 mcg x 4 — Inhaled Staccato Fentanyl, 25 mcg x 4 doses
  Arms: Inhaled fentanyl 25 mcg x 4
Drug: Inhaled Fentanyl 25 mcg x 6 — Inhaled Staccato Fentanyl, 25 mcg x 6 doses
  Arms: Inhaled fentanyl 25 mcg x 6
Drug: Inhaled Fentanyl 25 mcg x 12 — Inhaled Staccato Fentanyl, 25 mcg x 12 doses
  Arms: Inhaled fentanyl 25 mcg x 12

SUMMARY:
The Phase I clinical trial in approximately 50 healthy volunteers will be conducted at a single clinical center in two stages. Stage 1 is an open-label, cross-over comparison of a single dose of Staccato Fentanyl and an equivalent dose of intravenous (IV) fentanyl. Stage 2 is a randomized, doubleblind, placebo-controlled dose escalation of Staccato Fentanyl, evaluating multiple doses of fentanyl. The three primary aims of the Phase I clinical trial are to evaluate the pharmacokinetics (PK) and absolute bioavailability for Fentanyl, compare the Staccato Fentanyl PK profile to the IV fentanyl PK profile, and examine the tolerability and safety of Staccato Fentanyl in a non-opioid-tolerant, healthy volunteer population.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between the ages of 18 to 55 years, inclusive.
2. Subjects with a body mass index (BMI) ≥ 21 and ≤ 30.
3. Female subjects who are not pregnant, or are surgically sterile or 2 years postmenopausal. If of childbearing potential, she must be using a medically-accepted method of birth control and agree to continue use of this method for at least 30 days after the study (i.e., barrier method with spermicide, steroidal contraceptive [oral, transdermal, and implanted, including Depo-Provera; contraceptives must be used in conjunction with a barrier method], or intrauterine device).
4. Subjects who speak, read, and understand English and are willing and able to provide written informed consent on an IRB-approved form prior to the initiation of any study procedures.
5. Subjects who are willing and able to be confined to the Clinical Research Unit (CRU) for approximately 10 hours and comply with the study schedule and study requirements.
6. Subjects who are in good general health as determined by a complete medical history, physical examination, 12-lead ECG, spirometry, blood chemistry profile, hematology, and urinalysis.

Exclusion Criteria:

1. Subjects who regularly consume large amounts of xanthine-containing substances (i.e., more than 5 cups of coffee or equivalent amounts of xanthine-containing substances per day).
2. Subjects who have taken prescription or nonprescription medication (with the exception of vitamins, acetaminophen, and steroidal contraceptives for women of child-bearing potential if medically necessary) within 5 days of Visits 2 or 3.
3. Subjects who have had an acute illness within 5 days of either Visit 2 or 3.
4. Subjects who have received an investigational drug within 30 days (or within 5 half lives of the investigational drug) prior to Visit 2 or 3.
5. Subjects who have smoked tobacco within the last year.
6. Subjects who have a history within the past 2 years of drug or alcohol dependence or abuse as defined by DSM-4.
7. Subjects with a history of HIV positivity.
8. Subjects with a history of allergy or intolerance to opioids.
9. Subjects who test positive for alcohol or have a positive urine drug screen at any study visit.
10. Subjects who have hypotension (systolic blood pressure ≤90 mmHg, diastolic blood pressure ≤50 mmHg), or hypertension (systolic blood pressure ≥140 mmHg, diastolic blood pressure ≥90 mmHg).
11. Subjects who have a clinically significant ECG abnormality (beyond 1st degree heart block).
12. Subjects with a history of unstable angina, syncope, coronary artery disease, myocardial infarction, congestive heart failure (CHF), stroke, transient ischemic attack (TIA), or a significant neurological disorder.
13. Subjects who have a history of pulmonary disease (asthma, bronchitis, bronchospasm, emphysema).
14. Subjects who have an FEV1 less than 80% of predicted values on spirometry assessments at Visit 1.
15. Female subjects who are breastfeeding or have a positive pregnancy test at any visit must be excluded.
16. Subjects who have any other disease or condition, by history, physical examination, or laboratory abnormalities that in the investigator's opinion, would present undue risk to the subject, or may confound the interpretation of study results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2006-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To establish the plasma PK profile of fentanyl following single and multiple Staccato Fentanyl doses | 8 hours

SECONDARY OUTCOMES:
To assess Staccato Fentanyl absolute bioavailability and dose proportionality | 8 hours
Safety and Tolerability of Staccato Fentanyl | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tong J Gan, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Background] Macleod DB, Habib AS, Ikeda K, Spyker DA, Cassella JV, Ho KY, Gan TJ. Inhaled fentanyl aerosol in healthy volunteers: pharmacokinetics and pharmacodynamics. Anesth Analg. 2012 Nov;115(5):1071-7. doi: 10.1213/ANE.0b013e3182691898. Epub 2012 Sep 13. PMID 22984155